CLINICAL TRIAL: NCT04820959
Title: Validation of New Therapeutic Targets to Prevent Collagen Accumulation During Cardiac Fibrosis: Procollagen C-proteinase Enhancers
Acronym: CARDIACTIV
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Centre Hospitalier Universitaire Dijon (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: BOUCHOT ANR 2017
Record Dates: First submitted 2021-03-25; First posted 2021-03-29 (Actual); Last update posted 2024-02-28 (Actual); Status verified 2024-02

CONDITIONS: Valvulopathy; Heart Surgery; Procollagen C-Proteinase Enhancers
MeSH Terms: conditions — Heart Valve Diseases | interventions — Biopsy; Blood Specimen Collection

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Biological: Biopsies — Three endomyocardial intraoperative biopsies were performed on the left ventricle.
  Resection of the left atrium in the event of atrial fibrillation.
Biological: Blood sampling — Pre-operative blood sampling

SUMMARY:
Heart failure is characterized by cardiac fibrosis linked to extracellular collagen deposits. Collagens are synthesized as soluble precursors, procollagens, which must undergo proteolytic maturation to assemble into fibres. This step is under the control of two extracellular proteins, procollagen C-proteinase enhancer 1 and 2 (PCPE-1 and -2). The mechanism of action of these highly effective and specific activators was recently elucidated by one of our partners. Preliminary results, as well as data from the literature, indicate a strong correlation between the expression rates of PCPEs and cardiac fibrosis. The aim of this study is to validate in humans, by analysis of endomyocardial tissue biopsies, the hypothesis that PCPEs contribute to the anarchic accumulation of collagen during cardiac fibrosis and to evaluate the interest of developing new diagnostic and therapeutic strategies for cardiac fibrosis using PCPE agonists.

ELIGIBILITY:
Inclusion Criteria:

* Person who has given written consent
* Patient aged 18 to 85 for men and 60 to 85 for women
* Patient requiring cardiac surgery for aortic valve replacement or aortic plastic surgery or aortic plasty or ascending aorta replacement more or less associated with aortic valve surgery

Exclusion Criteria:

* Person not affiliated or not benefiting from national health insurance
* Person subject to a measure of legal protection (curatorship, guardianship)
* Person deprived of liberty, by judicial or administrative decision
* Major incapable or incapable of giving consent
* Minor
* Pregnant or breastfeeding woman
* Emergency Surgery
* Acute Infectious Endocarditis

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 66 (Actual)
Dates: Start 2020-10-04 (Actual); Primary Completion 2022-07-07 (Actual); Study Completion 2022-07-07 (Actual)

PRIMARY OUTCOMES:
Myocardial fibrosis rate | Through study completion, an average of 1 year
  Measurement of the level of myocardial fibrosis in myocardial tissue.
Rate of PCPE-1/2 | Through study completion, an average of 1 year
  Measurement of PCPE-1/2 rate in myocardial tissue.

CONTACTS AND LOCATIONS:
Locations (1):
- CHU Dijon Bourgogne, Dijon, France